CLINICAL TRIAL: NCT07324668
Title: The Effects of a Multiple Intervention Approach Applied to Postmenopausal Women on Quality of Life, Self-efficacy, and Urinary Incontinence Severity: a Temporal Analysis
Brief Title: Effects of Multiple Intervention on Postmenopausal Women With UI
Acronym: UI Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Şeyma SOYANIT ERASLAN, Dr., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-1075
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence; Postmenopausal
Keywords: Postmenopause; Women's health; Multimodal intervention; Urinary incontinence; Quality of life; Effectiveness
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups:
  1. Experimental Group 1 will perform Tai Chi and Kegel exercises 3 days per week,
  2. Experimental Group 2 will perform Tai Chi and Kegel exercises 6 days per week, and
  3. the Control Group will receive no intervention. All groups will be evaluated at baseline and after 8 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Tai Chi and Kegel, 3 days/week) (Experimental): articipants will perform Tai Chi and Kegel exercises 3 days per week for 8 weeks.
  Interventions: Behavioral: Combined Exercise Program
- Intervention Group 2 (Tai Chi and Kegel, 6 days/week) (Experimental): Participants will perform Tai Chi and Kegel exercises 6 days per week for 8 weeks.
  Interventions: Behavioral: Combined Exercise Program
- Control Group (No Intervention): Participants will receive no exercise or educational intervention and will continue their usual daily routines.

INTERVENTIONS:
Behavioral: Combined Exercise Program — Participants will receive education on urinary incontinence, Kegel and Tai Chi exercises, brochures and videos, and perform exercises 3 days/week for 8 weeks with reminders
  Arms: Intervention Group 1 (Tai Chi and Kegel, 3 days/week)
Behavioral: Combined Exercise Program — Participants will receive same education and materials as Group 1 and perform exercises 6 days/week for 8 weeks with reminders.
  Arms: Intervention Group 2 (Tai Chi and Kegel, 6 days/week)

SUMMARY:
Study

The purpose of this clinical trial was to investigate the effects of a multi-intervention approach, including Kegel and Tai Chi exercises, on quality of life, self-efficacy, and urinary incontinence severity in postmenopausal women.

Key Questions the Study Aims to Answer:

How does the multi-intervention approach affect quality of life?

Does the multi-intervention approach affect women's self-efficacy?

How does the multi-intervention approach affect urinary incontinence severity?

How does the frequency of exercises (3 days per week vs. 6 days per week) affect these outcomes?

Do the effects of the intervention change temporally over the 8-week period?

Who is Eligible?

Women aged 45 and over who have gone through menopause

Those who wish to volunteer for the study

Those who have no communication barriers

Those who have not previously received treatment for urinary incontinence

Those who can use a smartphone or WhatsApp

Those who experience urine leakage when coughing or sneezing

Study Application:

The exercises will be administered for 8 weeks.

Participants will be taught how to perform the exercises and will be demonstrated through brochures and videos.

Reminders will be provided during the exercises.

ELIGIBILITY:
Inclusion Criteria:

- Being female

Having undergone menopause

Willingness to participate in the study

No communication barriers

Not receiving any treatment for urinary incontinence

Owning a smartphone

Having WhatsApp installed

Experiencing urinary leakage when coughing or sneezing, according to the International Continence Society (ICS) definition

Exclusion Criteria:

Having communication barriers

Not being in menopause

Not owning a smartphone

Not experiencing urinary incontinence

Having received any treatment for urinary incontinence

Having undergone surgical menopause

-

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 117 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Urinary Incontinence Severity Measured by [İnkontinans Şiddet İndeksi] | 8 weeks (baseline and post-intervention)
  Quality of life related to urinary incontinence will be assessed using a validated questionnaire. Differences from baseline to post-test will be evaluated.

SECONDARY OUTCOMES:
Quality of Life Related to Urinary Incontinence | 8 weeks (baseline and post-intervention)
  Quality of life related to urinary incontinence will be assessed using a validated questionnaire. Differences from baseline to post-test will be evaluated.
Self-Efficacy in Managing Urinary Incontinence | Baseline and 8 weeks post-intervention
  Participants' self-efficacy will be measured using a validated scale, comparing baseline and post-test scores.

IPD SHARING:
Plan to Share IPD: Undecided